CLINICAL TRIAL: NCT00542204
Title: Patient-Centered Online Disease Management Using a Personal Health Record System
Brief Title: Use of Online Personalized Health Record System to Promote Self-Management of Diabetes
Acronym: EMPOWER-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Sutter Health (Other)
Responsible Party: Principal Investigator, Paul Tang, Vice President, Palo Alto Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS017179-01 (AHRQ)
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Blood Glucose Self-Monitoring; Home Blood Glucose Monitoring; Internet; Personal Health Record (PHR); Health Information Technology (HIT); Care management; Disease Management; Diabetes self-management; Consumer Health Information; Medical Records Systems, Computerized; Computerized Medical Records System; Automated Medical Records System; Electronic Health Record (EHR); Remote patient monitoring
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online disease management (Experimental): The PAMFOnline-mediated Personalized Health Care Program, which couples a multidisciplinary diabetes care management team with an EHR-integrated Online Disease Management (ODM) system.
  Interventions: Behavioral: Online disease management
- Usual care (No Intervention): Usual medical care. No access to the PHCP electronic system and self-management tools supporting this care management.

INTERVENTIONS:
Behavioral: Online disease management — The Personalized Health Care Program couples a multidisciplinary care management team with an EHR-integrated Online Disease Management (ODM) system.
  Other Names: EMPOWER-D
  Arms: Online disease management

SUMMARY:
Diabetes is a major, growing, and costly chronic disease in the U.S., and implementation of recommended diabetes care remains poor, not merely suboptimal, and varied for a sizable proportion of Americans with diabetes. To further reduce the treatment and adherence gaps in diabetes care, the researchers propose to evaluate a Customized, Continuous Care Management (CCCM) program that actively supports a partnership between the patient and his/her multidisciplinary care management (CM) team using an online disease management (ODM) system, which is integrated with a comprehensive electronic health record (EHR) system that includes a personal health record and secure patient-clinician messaging capabilities. The CCCM program builds upon CM strategies proven effective in past studies and creates an ODM system that is built upon and fully integrated with a leading, commercially available EHR product - providing a blueprint for instituting customized, continuous care management for many different chronic conditions in a range of ambulatory care settings.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Have a designated Palo Alto Medical Foundation Primary Care Provider (PCP)
* Seen in primary or specialty care at the Palo Alto Division at least once in the preceding 24 months
* Diagnosis of diabetes
* Baseline A1C >= 7.5%

Exclusion Criteria:

* Initial diagnosis of diabetes within the last 12 months
* Diagnosis of Type 1 diabetes
* Inability to speak and read in English
* Lack of regular access to a computer with Internet and email capabilities
* Unwilling to perform any self-monitoring at home, including blood glucose and blood pressure%
* Pregnant, planning to become pregnant, or lactating
* Currently enrolled in a care management program at Palo Alto Medical Foundation or elsewhere
* PCP determination that the study is inappropriate or unsafe for the patient
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | Baseline, 6 months and 12 months

SECONDARY OUTCOMES:
Self-management practices(e.g., medication adherence, home monitoring of glucose and BP, diet, and exercise) | Baseline, 6 months and 12 months
Processes of care (e.g., frequency of lab testing) | Baseline, 6 months and 12 months
Cardiovascular risk (e.g., blood pressure and lipids) | Baseline, 6 months and 12 months
Patient experience and satisfaction (e.g., relevant CAHPS measures) | Baseline and 12 months
Patient psychosocial well-being (e.g., diabetes-related emotional distress) | Baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tang, M.D., Principal Investigator — Palo Alto Medical Foundation
Locations (6):
- United States (6):
  - PAMF Palo Alto Health Care Division, Fremont, California
  - PAMF Palo Alto Health Care Division, Los Altos, California
  - PAMF Camino Region, Mountain View, California
  - PAMF Palo Alto Health Care Division, Palo Alto, California
  - PAMF Palo Alto Health Care Division, Redwood City, California
  - PAMF Santa Cruz Medical Clinic, Santa Cruz, California

REFERENCES:
- [Derived] Tang PC, Overhage JM, Chan AS, Brown NL, Aghighi B, Entwistle MP, Hui SL, Hyde SM, Klieman LH, Mitchell CJ, Perkins AJ, Qureshi LS, Waltimyer TA, Winters LJ, Young CY. Online disease management of diabetes: engaging and motivating patients online with enhanced resources-diabetes (EMPOWER-D), a randomized controlled trial. J Am Med Inform Assoc. 2013 May 1;20(3):526-34. doi: 10.1136/amiajnl-2012-001263. Epub 2012 Nov 20. PMID 23171659